CLINICAL TRIAL: NCT05269966
Title: A Real-world, Prospective, Multi-center, Open-label, Phase IV Clinical Study to Evaluate the Safety and Effectiveness of Intravitreal Injections (IVI) of Brolucizumab in Patients With Neovascular Age-related Macular Degeneration (nAMD)
Brief Title: Study to Evaluate the Safety and Effectiveness of Intravitreal Injections (IVI) of Brolucizumab in Patients With Neovascular Age-related Macular Degeneration (nAMD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRTH258AIN01
Record Dates: First submitted 2022-02-16; First posted 2022-03-08 (Actual); Results first posted 2024-12-10 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Neovascular Age-related Macular Degeneration (nAMD)
Keywords: Macular degeneration; age-related macular degeneration (ARMD); vision loss; macula damage; retina damage; dry macular degeneration; wet macular degeneration; Subfoveal choroidal neovascularization (CNV) secondary to age-related macular degeneration; AMD; neovascular age-related macular degeneration; nAMD; retinal vein occlusion; RVO
MeSH Terms: conditions — Macular Degeneration; Vision Disorders; Geographic Atrophy; Wet Macular Degeneration; Choroidal Neovascularization; Retinal Vein Occlusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Brolucizumab (Experimental): Brolucizumab, formerly known as ESBA1008, is a humanized single-chain Fv (scFv) antibody fragment.
  Brolucizumab 6 mg was administered by Intravitreal (IVT) injections as per the Prescribing information (PI) and in line with the treating physician's clinical judgement. Patients received loading doses of brolucizumab at Day 0/Visit 1, Week 4/Visit 2 and Week 8/Visit 3. After the loading doses, at Week 16, disease activity assessment (DAA) was performed based on Best Corrected Visual Acuity (BCVA) and Optical Coherence Tomography (OCT) to assess whether the patient required q8w or q12w dosing.
  Interventions: Biological: Injection Brolucizumab

INTERVENTIONS:
Biological: Injection Brolucizumab — Single-chain antibody fragment (scFv)
  Brolucizumab 6 mg was administered by Intravitreal (IVT) injection as per the Prescribing information (PI) and in line with the treating physician's clinical judgement. Patients received loading doses of brolucizumab at Day 0/Visit 1, Week 4/Visit 2 and Week 8/Visit 3. After the loading doses, at Week 16, disease activity assessment (DAA) were performed based on Best Corrected Visual Acuity (BCVA) and Optical Coherence Tomography (OCT) to assess whether the patient required q8w or q12w dosing.
  Other Names: Trade Names: Pagenax, Beovu, Vsiqq

SUMMARY:
The purpose of this study was to generate additional safety and effectiveness data in Indian neovascular age-related macular degeneration (nAMD) patients that more closely resemble the real-world population intended to be treated with brolucizumab. This study was conducted as part of the post-marketing regulatory commitment to the Indian Health authority.

DETAILED DESCRIPTION:
The study was a prospective, multi-center, open-label, interventional phase IV clinical study.

The study treatment, i.e., brolucizumab was prescribed in terms of the marketing authorization; the assignment of the patient to the therapy was decided within the current practice and the medical indication. It was clearly separated from the decision to include the patient in the study.

All patients with Neovascular Age-related Macular Degeneration (nAMD) who were planned to be treated with brolucizumab and had provided informed consent were enrolled in the study. A total of 12 sites in India were evaluated for the study conduct. This is to note that site #03 was not selected, and site #07 was not initiated, and patients were enrolled in the study only from 10 sites.

The treatment period for each patient was 56 weeks after the start of brolucizumab treatment.

Study visits were scheduled at Week 4, Week 8, Week 16, and thereafter at intervals of 8 weeks or 12 weeks after disease activity assessment at Week 16. If the investigators required more frequent follow-up visits, it was done according to their discretion and clinical judgment. Any patient who suffered from IOI during the study period was not re-challenged with brolucizumab.

The study population consisted of adult male and female outpatients aged 50 years and above, diagnosed with nAMD for whom the treating the physician (Investigator) had prescribed treatment with brolucizumab 6 mg injection in adherence with the local Summary of Product Characteristics (SmPC) or Prescribing Information (PI).

ELIGIBILITY:
Inclusion Criteria:

* Female or male, treatment naïve patient with ≥50 years of age, with neovascular age-related macular degeneration (nAMD).
* Patient or legally acceptable representative (LAR) willing to voluntarily provide signed informed consent for participation in the study.

Note: In case where both eyes are affected, data of only one eye ['study eye'] will be recorded. Selection of the eye to be considered for the purpose of the study [referred to as 'study eye'] will be as per the Investigator's discretion.

Exclusion Criteria:

* Patients fulfilling any of the following criteria are not eligible for this study:
* Patient having other eye diseases that could compromise the VA.
* Patient with existing or suspected ocular or periocular infection in the study eye.
* Patient with an existing intraocular inflammation (IOI).
* Patient with uncontrolled glaucoma defined as intraocular pressure > 25 mmHg despite treatment with anti-glaucoma medication, or according to Investigator's judgment.
* Patient who has undergone intraocular surgery within 3 months prior to enrollment in this study.
* Patient having scar, fibrosis and atrophy involving the center of the fovea in the study eye.

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2022-03-09 (Actual); Primary Completion 2023-08-29 (Actual); Study Completion 2023-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (10):
- India (10):
  - Novartis Investigative Site, Asarwa, Ahmedabad
  - Novartis Investigative Site, Ahmedabad, Gujarat
  - Novartis Investigative Site, Bangalore, Karnataka
  - Novartis Investigative Site, Chennai, Tamil Nadu
  - Novartis Investigative Site, Hyderabad, Telangana
  - Novartis Investigative Site, Varanasi, Uttar Pradesh
  - Novartis Investigative Site, Kolkata, West Bengal
  - Novartis Investigative Site, Chandigarh
  - Novartis Investigative Site, Hugli
  - Novartis Investigative Site, New Delhi

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on https://www.clinicalstudydatarequest.com/.
URL: https://www.clinicalstudydatarequest.com/

REFERENCES:
- [Result] Rein DB, Wittenborn JS, Zhang X, Honeycutt AA, Lesesne SB, Saaddine J; Vision Health Cost-Effectiveness Study Group. Forecasting age-related macular degeneration through the year 2050: the potential impact of new treatments. Arch Ophthalmol. 2009 Apr;127(4):533-40. doi: 10.1001/archophthalmol.2009.58. PMID 19365036
- [Result] Kawasaki R, Yasuda M, Song SJ, Chen SJ, Jonas JB, Wang JJ, Mitchell P, Wong TY. The prevalence of age-related macular degeneration in Asians: a systematic review and meta-analysis. Ophthalmology. 2010 May;117(5):921-7. doi: 10.1016/j.ophtha.2009.10.007. Epub 2010 Jan 27. PMID 20110127
- [Result] Smith W, Assink J, Klein R, Mitchell P, Klaver CC, Klein BE, Hofman A, Jensen S, Wang JJ, de Jong PT. Risk factors for age-related macular degeneration: Pooled findings from three continents. Ophthalmology. 2001 Apr;108(4):697-704. doi: 10.1016/s0161-6420(00)00580-7. PMID 11297486
- [Result] Miller JW. Age-related macular degeneration revisited--piecing the puzzle: the LXIX Edward Jackson memorial lecture. Am J Ophthalmol. 2013 Jan;155(1):1-35.e13. doi: 10.1016/j.ajo.2012.10.018. PMID 23245386
- [Result] Ferris FL 3rd, Fine SL, Hyman L. Age-related macular degeneration and blindness due to neovascular maculopathy. Arch Ophthalmol. 1984 Nov;102(11):1640-2. doi: 10.1001/archopht.1984.01040031330019. PMID 6208888
- [Result] Lim LS, Mitchell P, Seddon JM, Holz FG, Wong TY. Age-related macular degeneration. Lancet. 2012 May 5;379(9827):1728-38. doi: 10.1016/S0140-6736(12)60282-7. PMID 22559899
- [Result] Shah AR, Del Priore LV. Progressive visual loss in subfoveal exudation in age-related macular degeneration: a meta-analysis using Lineweaver-Burke plots. Am J Ophthalmol. 2007 Jan;143(1):83-89. doi: 10.1016/j.ajo.2006.09.043. Epub 2006 Oct 20. PMID 17188044
- [Result] Shah AR, Del Priore LV. Natural history of predominantly classic, minimally classic, and occult subgroups in exudative age-related macular degeneration. Ophthalmology. 2009 Oct;116(10):1901-7. doi: 10.1016/j.ophtha.2009.03.055. Epub 2009 Jul 9. PMID 19592101
- [Result] Blinder KJ, Bradley S, Bressler NM, Bressler SB, Donati G, Hao Y, Ma C, Menchini U, Miller J, Potter MJ, Pournaras C, Reaves A, Rosenfeld PJ, Strong HA, Stur M, Su XY, Virgili G; Treatment of Age-related Macular Degeneration with Photodynamic Therapy study group; Verteporfin in Photodynamic Therapy study group. Effect of lesion size, visual acuity, and lesion composition on visual acuity change with and without verteporfin therapy for choroidal neovascularization secondary to age-related macular degeneration: TAP and VIP report no. 1. Am J Ophthalmol. 2003 Sep;136(3):407-18. doi: 10.1016/s0002-9394(03)00223-x. PMID 12967792
- [Result] Sommer A, Tielsch JM, Katz J, Quigley HA, Gottsch JD, Javitt JC, Martone JF, Royall RM, Witt KA, Ezrine S. Racial differences in the cause-specific prevalence of blindness in east Baltimore. N Engl J Med. 1991 Nov 14;325(20):1412-7. doi: 10.1056/NEJM199111143252004. PMID 1922252
- [Result] Wong TY, Chakravarthy U, Klein R, Mitchell P, Zlateva G, Buggage R, Fahrbach K, Probst C, Sledge I. The natural history and prognosis of neovascular age-related macular degeneration: a systematic review of the literature and meta-analysis. Ophthalmology. 2008 Jan;115(1):116-26. doi: 10.1016/j.ophtha.2007.03.008. Epub 2007 Aug 6. PMID 17675159
- [Result] Menrad A, Anderer FA. Expression of LDL receptor on tumor cells induced by growth factors. Anticancer Res. 1991 Jan-Feb;11(1):385-90. PMID 1850220
- [Result] Campbell JP, Bressler SB, Bressler NM. Impact of availability of anti-vascular endothelial growth factor therapy on visual impairment and blindness due to neovascular age-related macular degeneration. Arch Ophthalmol. 2012 Jun;130(6):794-5. doi: 10.1001/archophthalmol.2011.2480. No abstract available. PMID 22801846
- [Result] Bloch SB, Larsen M, Munch IC. Incidence of legal blindness from age-related macular degeneration in denmark: year 2000 to 2010. Am J Ophthalmol. 2012 Feb;153(2):209-213.e2. doi: 10.1016/j.ajo.2011.10.016. PMID 22264944
- [Result] Nguyen QD, Das A, Do DV, Dugel PU, Gomes A, Holz FG, Koh A, Pan CK, Sepah YJ, Patel N, MacLeod H, Maurer P. Brolucizumab: Evolution through Preclinical and Clinical Studies and the Implications for the Management of Neovascular Age-Related Macular Degeneration. Ophthalmology. 2020 Jul;127(7):963-976. doi: 10.1016/j.ophtha.2019.12.031. Epub 2020 Jan 17. PMID 32107066
- [Result] Dugel PU, Koh A, Ogura Y, Jaffe GJ, Schmidt-Erfurth U, Brown DM, Gomes AV, Warburton J, Weichselberger A, Holz FG; HAWK and HARRIER Study Investigators. HAWK and HARRIER: Phase 3, Multicenter, Randomized, Double-Masked Trials of Brolucizumab for Neovascular Age-Related Macular Degeneration. Ophthalmology. 2020 Jan;127(1):72-84. doi: 10.1016/j.ophtha.2019.04.017. Epub 2019 Apr 12. PMID 30986442
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2191

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In case where both eyes were affected, data of only one eye ['study eye'] was recorded. Selection of the eye to be considered for the purpose of the study [referred to as 'study eye'] was as per the Investigator's discretion.
Period: Overall Study
Arm/Group | Brolucizumab
Started | 105
Completed | 95
Not Completed | 10
Not completed — Adverse Event | 4
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 4
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Brolucizumab
Number analyzed (Participants) | 105
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.7 (9.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 63
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 105
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 105
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Incidence and Characteristics of Treatment-emergent Adverse Events During the 56 Weeks of Treatment With Brolucizumab.
Description: An adverse event (AE) is any untoward medical occurrence (e.g. any unfavorable and unintended sign [including abnormal laboratory findings], symptom or disease) in a clinical investigation participant after providing written informed consent for participation in the study.
  Treatment-emergent Adverse Events (TEAEs) in this study are defined as AEs suspected to be related to the study drug.
Time Frame: Adverse events were reported from first dose of study treatment until Week 48, plus 8 weeks follow up, to a maximum timeframe of 56 weeks.
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab
Number analyzed (Participants) | 105
Participants
  At least one AE | 67
  At least one Ocular AEs | 50
  At least one Ocular AE in the Study eye | 45
  At least one Ocular AE in the Fellow eye | 9
  Systemic (non-ocular) AEs | 31
  TEAEs | 3
  AEs related to brolucizumab | 3
  Ongoing AEs | 10
  CTCAE grade of AEs - Total | 67
  CTCAE grade of AEs - Mild | 63
  CTCAE grade of AEs - Moderate | 6
  CTCAE grade of AEs - Severe | 1
  CTCAE grade of AEs - Life Threatening | 0
  CTCAE grade of AEs - Death Related to AE | 0
  Serious adverse event | 0
  Serious AEs related to brolucizumab | 0
  AEs Action Taken - Total | 67
  AEs Action Taken - No action taken | 66
  AEs Action Taken - Investigational treatment permanently discontinued due to this adverse event | 5
  Outcome of AEs - Total | 67
  Outcome of AEs - Not Recovered or Not Resolved | 10
  Outcome of AEs - Recovered or resolved | 61
  Outcome of AEs - Recovering or resolving | 0
  Outcome of AEs - Recovered or resolved with sequelae | 0
  Outcome of AEs - Fatal | 0
  Outcome of AEs - Unknown | 0
  AEs leading to discontinuation from the study | 4
  AEs leading to death | 0
  Related AEs leading to death | 0

2. Secondary Outcome: Mean Change in Best-Corrected Visual Acuity (BCVA) From Baseline at Week 16 and Week 56 as Measured by Early Treatment Diabetic Retinopathy Study (ETDRS) Letters - Study Eye
Description: BCVA was assessed using Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing charts.
  Visual Function of the study eye was assessed using the ETDRS protocol.
  Min and max possible scores are 0-100 respectively. A higher score represents better visual functioning.
Time Frame: Baseline, Week 16, Week 56
Population: Full analysis set - The full analysis set (FAS) comprises all patients who received at least one IVT injection of study treatment without protocol deviation with impact and with an assessment at the specified timeframe.
Measure: Mean (Standard Deviation); unit: Letters read
Arm/Group | Brolucizumab
Number analyzed (Participants) | 81
Letters read
  Week 16 | 10.7 (12.53)
  Week 56 | 15.3 (13.74)

3. Secondary Outcome: Change in Best-Corrected Visual Acuity (BCVA) From Baseline at Week 16 and Week 56 as Measured by Early Treatment Diabetic Retinopathy Study (ETDRS) Letters - Median - Study Eye
Description: as for outcome 2
Time Frame: Baseline, Week 16, Week 56
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Letters read
Arm/Group | Brolucizumab
Number analyzed (Participants) | 81
Letters read
  Week 16 | 7.0 [-16 to 70]
  Week 56 | 15.0 [-29 to 70]

4. Secondary Outcome: Number and Percentage (%) of Participants With Gain in Best-Corrected Visual Acuity (BCVA) of 15/10/5 ETDRS Letters or More From Baseline at Week 16 and Week 56 - Study Eye
Description: as for outcome 2
Time Frame: Baseline, Week 16 and Week 56
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab
Number analyzed (Participants) | 105
Participants
  Week 16 - Total Visual Acuity Score (ETDRS letters) Gain ≥ 15 ETDRS letters | 27 [17.68 to 35.17]
  Week 16 -Total Visual Acuity Score (ETDRS letters) Gain ≥ 10 ETDRS letters | 41 [29.67 to 49.06]
  Week 16 -Total Visual Acuity Score (ETDRS letters) Gain ≥ 5 ETDRS letters | 79 [65.86 to 83.14]
  Week 56 - Total Visual Acuity Score (ETDRS letters) Gain ≥ 15 ETDRS letters | 46 [34.14 to 53.83]
  Week 56 - Total Visual Acuity Score (ETDRS letters) Gain ≥ 10 ETDRS letters | 62 [49.02 to 68.55]
  Week 56 - Total Visual Acuity Score (ETDRS letters) Gain ≥ 5 ETDRS letters | 78 [64.83 to 82.32]

5. Secondary Outcome: Number and Percentage (%) of Participants With Loss in Best-Corrected Visual Acuity (BCVA) of 15/10/5 ETDRS Letters or More From Baseline at Week 16 and Week 56 - Study Eye
Description: as for outcome 2
Time Frame: Baseline, Week 16 and Week 56
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab
Number analyzed (Participants) | 105
Participants
  Week 16 - Total Visual Acuity Score (ETDRS letters) loss ≥ 15 ETDRS letters | 2
  Week 16 -Total Visual Acuity Score (ETDRS letters) loss ≥ 10 ETDRS letters | 2
  Week 16 -Total Visual Acuity Score (ETDRS letters) loss ≥ 5 ETDRS letters | 3
  Week 56 - Total Visual Acuity Score (ETDRS letters) loss ≥ 15 ETDRS letters | 2
  Week 56 - Total Visual Acuity Score (ETDRS letters) loss ≥ 10 ETDRS letters | 2
  Week 56 - Total Visual Acuity Score (ETDRS letters) loss ≥ 5 ETDRS letters | 3

6. Secondary Outcome: Number of Anti-VEGF Injections, During the 56 Weeks of Treatment With Brolucizumab - Study Eye
Description: Characterize the number of anti-VEGF injections during the 56 weeks of treatment with brolucizumab.
Time Frame: Week 56
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: Injections
Arm/Group | Brolucizumab
Number analyzed (Participants) | 105
Injections | 6.2 (1.30)

7. Secondary Outcome: Number of Non-injection Visits During the 56 Weeks of Treatment With Brolucizumab
Description: Characterize number of non-injection visits during the 56 weeks of treatment with brolucizumab.
Time Frame: Week 56
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: Visits
Arm/Group | Brolucizumab
Number analyzed (Participants) | 105
Visits | 0.2 (0.71)

8. Secondary Outcome: Total Number of Visits During the 56 Weeks of Treatment With Brolucizumab.
Description: Characterize the total number of visits during the 56 weeks of treatment with brolucizumab.
Time Frame: Week 56
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: visits
Arm/Group | Brolucizumab
Number analyzed (Participants) | 105
visits | 6.2 (1.30)

9. Secondary Outcome: Number and Percentage (%) of Participants With at Least One Duration of Interval Between Injections ≥ 8 Weeks But <12 Weeks.
Time Frame: Week 56
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab
Number analyzed (Participants) | 105
Participants | 27

10. Secondary Outcome: Number and Percentage (%) of Participants With at Least One Duration of Interval Between Injections ≥ 12 Weeks.
Time Frame: Week 56
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab
Number analyzed (Participants) | 105
Participants
  At least one duration of interval between injections ≥ 12 weeks | 74
  q8w dosing | 27
  q12w dosing | 74

11. Secondary Outcome: Number and Percentage (%) of Participants With Absence of Intra-retinal Fluid (IRF) From Baseline to Week 16 and Week 56 - for Patients Where IRF Was Absent at Baseline - Study Eye
Description: Estimate effect of brolucizumab on fluid (increased/reduced/unchanged) from baseline to week 16 and week 56 based on Optical Coherence Tomography (SD-OCT) Image Analysis from the central reading center.
Time Frame: Week 16 and Week 56
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab
Number analyzed (Participants) | 105
Participants
  Week 16 Absent | 2
  Week 16 Decreased | 0
  Week 16 Increased | 0
  Week 56 Absent | 2
  Week 56 Decreased | 0
  Week 56 Increased | 0

12. Secondary Outcome: Number and Percentage (%) of Participants With Absence of Intra-retinal Fluid (IRF) From Baseline to Week 16 and Week 56 - for Patients Where IRF Was Present at Baseline - Study Eye
Description: as for outcome 11
Time Frame: Week 16 and Week 56
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab
Number analyzed (Participants) | 105
Participants
  Week 16 Absent | 23
  Week 16 Decreased | 54
  Week 16 Increased | 22
  Week 56 Absent | 43
  Week 56 Decreased | 50
  Week 56 Increased | 7

13. Secondary Outcome: Number and Percentage (%) of Participants With Absence of Sub-retinal Fluid (SRF) From Baseline to Week 16 and Week 56 - for Patients Where SRF Was Absent at Baseline - Study Eye
Description: Estimate effect of brolucizumab on fluid from baseline to week 16 and week 56. Assessed by Spectral domain optical coherence tomography (SD-OCT) from the central reading center.
Time Frame: Week 16 and Week 56
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab
Number analyzed (Participants) | 105
Participants
  Week 16 Absent | 10
  Week 16 Decreased | 0
  Week 16 Increased | 0
  Week 56 Absent | 11
  Week 56 Decreased | 0
  Week 56 Increased | 0

14. Secondary Outcome: Number and Percentage (%) of Participants With Absence of Sub-retinal Fluid (SRF) From Baseline to Week 16 and Week 56 - for Patients Where SRF Was Present at Baseline - Study Eye
Description: as for outcome 13
Time Frame: Week 16 and Week 56
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab
Number analyzed (Participants) | 105
Participants
  Week 16 Absent | 20
  Week 16 Decreased | 57
  Week 16 Increased | 14
  Week 56 Absent | 30
  Week 56 Decreased | 57
  Week 56 Increased | 4

15. Secondary Outcome: Estimate CST Change From Baseline at Week 16 and Week 56 - Mean - Study Eye
Description: Estimate effect of brolucizumab on central subfield thickness (CST) from baseline to week 16 and week 56 as measured by Optical Coherence Tomography (in µm).
Time Frame: Baseline, Week 16 and Week 56
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: μm
Arm/Group | Brolucizumab
Number analyzed (Participants) | 105
μm
  Week 16 | -106.9 (129.14)
  Week 56 | -103.1 (152.64)

16. Primary Outcome: Incidence of Treatment-emergent Adverse Events During the 56 Weeks of Treatment With Brolucizumab - Ocular AEs - Preferred Term
Description: as for outcome 1
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab
Number analyzed (Participants) | 105
Participants
  Patients with at least one TEAE | 3
  Eye disorders - Total | 3
  Eye disorders - Vitritis | 2
  Eye disorders - Retinal vasculitis | 1
  Eye disorders - Uveitis | 1

17. Primary Outcome: Characteristics of Treatment-emergent Adverse Events During the 56 Weeks of Treatment With Brolucizumab
Description: as for outcome 1
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab
Number analyzed (Participants) | 105
Participants
  TEAEs | 3
  Ocular AEs | 3
  Systemic (non-ocular) AEs | 0
  Suspected TEAEs related to the study medication | 3
  Serious TEAEs | 0
  TEAEs leading to death | 0
  TEAEs leading to discontinuation of study | 2

18. Primary Outcome: Incidence of Ocular Adverse Event (AEs) by System Organ Class (SOC) and Preferred Term (PT) During the 56 Weeks of Treatment With Brolucizumab
Description: An adverse event (AE) is any untoward medical occurrence (e.g. any unfavorable and unintended sign [including abnormal laboratory findings], symptom or disease) in a clinical investigation participant after providing written informed consent for participation in the study.
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab
Number analyzed (Participants) | 105
Participants
  Patients with at least one Ocular AEs | 50
  Eye disorders - Total | 48
  Eye disorders - Conjunctival hemorrhage | 13
  Eye disorders - Cataract | 10
  Eye disorders - Vision blurred | 9
  Eye disorders - Ocular hyperemia | 7
  Eye disorders -Lacrimation increased | 6
  Eye disorders - Eye pain | 4
  Eye disorders - Eye pruritus | 4
  Eye disorders - Visual impairment | 3
  Eye disorders - Macular scar | 2
  Eye disorders - Retinal hemorrhage | 2
  Eye disorders -Vitritis | 2
  Eye disorders - Conjunctival hyperemia | 1
  Eye disorders - Eye irritation | 1
  Eye disorders - Retinal pigment epithelial tear | 1
  Eye disorders - Retinal vasculitis | 1
  Eye disorders - Swelling of eyelid | 1
  Eye disorders -Uveitis | 1
  Eye disorders - Vitreous floaters | 1
  Surgical and medical procedures - Cataract operation | 6
  General disorders and administration site conditions - Total | 3
  General disorders and administration site conditions -Injection site pain | 1
  General disorders and administration site conditions - Instillation site lacrimation | 1
  General disorders and administration site conditions -Sensation of foreign body | 1
  Infections and infestations - Conjunctivitis | 1

19. Secondary Outcome: Estimate CST Change From Baseline at Week 16 and Week 56 - Median - Study Eye
Description: as for outcome 15
Time Frame: Baseline, Week 16 and Week 56
Population: Full analysis set
Measure: Median (Inter-Quartile Range); unit: μm
Arm/Group | Brolucizumab
Number analyzed (Participants) | 105
μm
  Week 16 | -60.0 [-923 to 84]
  Week 56 | -66.5 [-902 to 369]

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment until Week 48, plus 8 weeks follow up, to a maximum timeframe of 56 weeks.
Arm/Group | Brolucizumab
All-Cause Mortality (participants affected / at risk) | 0/105
Serious Adverse Events (participants affected / at risk) | 0/105
Other Adverse Events (participants affected / at risk) | 67/105
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brolucizumab (N=105)
Cataract- Fellow eye (Eye disorders) | 4
Cataract- Study eye (Eye disorders) | 8
Conjunctival haemorrhage- Study eye (Eye disorders) | 13
Conjunctival hyperaemia- Study eye (Eye disorders) | 1
Eye irritation- Study eye (Eye disorders) | 1
Eye pain- Study eye (Eye disorders) | 4
Eye pruritus- Study eye (Eye disorders) | 4
Lacrimation increased- Fellow eye (Eye disorders) | 2
Lacrimation increased- Study eye (Eye disorders) | 4
Macular scar- Study eye (Eye disorders) | 2
Ocular hyperaemia- Study eye (Eye disorders) | 7
Retinal haemorrhage- Study eye (Eye disorders) | 2
Retinal pigment epithelial tear- Study eye (Eye disorders) | 1
Retinal vasculitis- Study eye (Eye disorders) | 1
Swelling of eyelid- Study eye (Eye disorders) | 1
Uveitis- Study eye (Eye disorders) | 1
Vision blurred- Fellow eye (Eye disorders) | 4
Vision blurred- Study eye (Eye disorders) | 6
Visual impairment- Study eye (Eye disorders) | 3
Vitreous floaters- Study eye (Eye disorders) | 1
Vitritis- Study eye (Eye disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Asthenia (General disorders) | 1
Injection site pain- Study eye (General disorders) | 1
Instillation site lacrimation- Study eye (General disorders) | 1
Pain (General disorders) | 1
Pyrexia (General disorders) | 13
Sensation of foreign body- Fellow eye (General disorders) | 1
Conjunctivitis- Study eye (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Blood pressure increased (Investigations) | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Erythema (Skin and subcutaneous tissue disorders) | 2
Cataract operation- Fellow eye (Surgical and medical procedures) | 3
Cataract operation- Study eye (Surgical and medical procedures) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-05-06): https://cdn.clinicaltrials.gov/large-docs/66/NCT05269966/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-16): https://cdn.clinicaltrials.gov/large-docs/66/NCT05269966/SAP_001.pdf